CLINICAL TRIAL: NCT01990573
Title: Methadone in Pediatric Anesthesia II
Brief Title: Methadone in Pediatric Anesthesiology II
Acronym: MEPAII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201302099
Record Dates: First submitted 2013-11-07; First posted 2013-11-21 (Estimated); Results first posted 2020-01-28 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Pain
Keywords: spinal surgery; Methadone
MeSH Terms: conditions — Pain | interventions — Amidines; Methadone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- methadone HCl 0.3 mg/kg (Experimental): 0.3mg/kg IV methadone HCl
  Interventions: Drug: 0.3mg/kg IV methadone HCl
- methadone HCl 0.4 mg/kg (Experimental): 0.4mg/kg IV methadon HCl
  Interventions: Drug: 0.4mg/kg IV methadon HCl
- control group (Active Comparator): control no methadone, standard of care opioids.
  Interventions: Other: control no methadone

INTERVENTIONS:
Drug: 0.3mg/kg IV methadone HCl — Group I will receive 0.3mg/kg IV methadone HCl
  Other Names: methadone HCl, dolophine
  Arms: methadone HCl 0.3 mg/kg
Drug: 0.4mg/kg IV methadon HCl — Group II will receive 0.4mg/kg IV methadone HCl.
  Other Names: methadone HCl, dolophine
  Arms: methadone HCl 0.4 mg/kg
Other: control no methadone — The control group will not receive methadone.
  Arms: control group

SUMMARY:
Three arm randomized controlled trial to evaluate the efficacy of a single dose of intraoperative methadone in reducing post-operative pain and opioid consumption in adolescents undergoing posterior spinal fusion. Our secondary goal is to determine the pharmacokinetics of IV methadone in children (0.3 and 0.4 mg/kg).

DETAILED DESCRIPTION:
Randomized, controlled, modified dose-escalation design. Patients receive standard monitoring for anesthesia and postoperative care. Surgical and anesthesia (except for opioid use) care are not altered for study purposes. All patients are induced by propofol and muscle relaxants. In the first cohort (n=30 evaluable), subjects are randomized 1:2 to either control (standard intraop opioid at anesthesiologists' discretion) or methadone HCl (0.4 mg/kg ideal body weight, IBW). In the second cohort (n=30 evaluable), subjects are randomized 1:2 to either control (standard intraop opioid) or methadone HCl (0.3 mg/kg ideal body weight, IBW). Subjects in the study groups will receive methadone (IV bolus, after induction of anesthesia) as their primary intraoperative opioid, rather than leaving the choice of intraoperative opioid to the anesthesiologist. Intraoperative breakthrough pain will be treated at the discretion of the anesthesiologist with fentanyl. In the control groups, intraoperative opioid administration will be left at the discretion of the anesthesia providers. Patient controlled analgesia as prescribed by the clinical team, using hydromorphone or morphine, will be used to treat postoperative pain relief.

ELIGIBILITY:
Inclusion Criteria.

* Age 11-18 years
* Undergoing general anesthesia and idiopathic posterior spinal surgery with anticipated postop inpatient stay of > 3 days
* Signed, written, informed consent from legal guardians and assent from patient

Exclusion Criteria.

* History of or known liver or kidney disease.
* Females who are pregnant or nursing.
* Children with developmental delay
* Children undergoing surgery for scoliosis of musculoskeletal origin

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 51 (Actual)
Dates: Start 2013-04-10 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anshuman Sharma, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 53 signed consents however, 2 participants withdrew prior to randomization:
  1 per family request
  1 unable to complete
Period: Overall Study
Arm/Group | Methadone HCl 0.3 mg/kg | Methadone HCl 0.4 mg/kg | Control Group
Started | 20 | 14 | 17
Completed | 20 | 14 | 16
Not Completed | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Methadone 0.3 mg/kg: 0.3mg/kg IV methadone
  0.3mg/kg IV methadone : Group I will receive 0.3mg/kg IV methadone
- Methadone 0.4 mg/kg: 0.4mg/kg IV methadone
  0.4mg/kg IV methadone: Group II will receive 0.4mg/kg IV methadone .
- Total: Total of all reporting groups
Arm/Group | Methadone 0.3 mg/kg | Methadone 0.4 mg/kg | Control Group | Total
Number analyzed (Participants) | 20 | 14 | 17 | 51
Age, Continuous [Mean (Standard Deviation); unit: Years] | 13.7 (1.5) | 14.8 (1.9) | 14.5 (1.9) | 14.3 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 11 | 10 | 35
  Male | 6 | 3 | 7 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 18 | 12 | 14 | 44
  Other | 2 | 2 | 3 | 7
Region of Enrollment [Number; unit: participants]
  United States | 20 | 14 | 17 | 51
American Society of Anesthesiologists (ASA) Physical Satus [Count of Participants; unit: Participants] — The purpose of the system is to assess and communicate a patient's pre-anesthesia medical co-morbidities. The classification system alone does not predict the perioperative risks, but used with other factors (eg, type of surgery, frailty, level of deconditioning), it can be helpful in predicting perioperative risks.
  Participants
    ASA 1 -A normal healthy patient | 16 | 6 | 6 | 28
    ASA 2 - A patient with mild systemic disease | 4 | 8 | 11 | 23
Pre-operative pain score [Mean (Standard Deviation); unit: units on a scale] — Numeric Pain Score was used to measure patient reported pain. The scale, previously validated, measures pain from 0 to 10, zero being no pain and 10 being the highest imaginable pain
  units on a scale | 1.6 (2.1) | .6 (1.2) | 1.9 (3.1) | 1.4 (2.3)
Expected Post-operative Pain Score [Mean (Standard Deviation); unit: 0-10 units on a Visual Analog scale] — Numeric Pain Score was used to measure patient reported pain. The scale, previously validated, measures pain from 0 to 10, zero being no pain and 10 being the highest imaginable pain
  0-10 units on a Visual Analog scale | 7.9 (2.1) | 6.9 (2.0) | 7.5 (1.9) | 7.2 (2.0)
BMI [Mean (Standard Deviation); unit: kg/m^2 scale] | 21.6 (3.8) | 21.3 (2.4) | 22.4 (4.8) | 21.7 (3.8)

OUTCOME MEASURES:

1. Primary Outcome: Total Opioid Consumption (Morphine Equivalent)
Description: Measure of overall morphine consumption
Time Frame: 6 days
Measure: Mean (Standard Deviation); unit: mg/kg
Arm/Group | Methadone HCl 0.3 mg/kg | Methadone HCl 0.4 mg/kg | Control Group
Number analyzed (Participants) | 20 | 14 | 16
mg/kg | 2.22 (.84) | 2.37 (.86) | 3.28 (.93)
Statistical Analysis 1: Comparison: Methadone HCl 0.3 mg/kg vs Methadone HCl 0.4 mg/kg vs Control Group; Test type: Other — ANOVA; p = .002, ANOVA; F statistic = .002

2. Primary Outcome: Pain Scores
Description: Assessments are made in the postoperative period by a trained member of the research team blinded to intraoperative use of methadone. These will be conducted on each post-operative day until discharge or post op day 6, whichever comes first. Pain intensity is assessed using the numeric pain score (0-10) scale employed by the inpatient nursing staff and previously validated .
Time Frame: 6 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Methadone HCl 0.3 mg/kg | Methadone HCl 0.4 mg/kg | Control Group
Number analyzed (Participants) | 20 | 14 | 16
score on a scale | 4.7 (2.4) | 4.6 (2.9) | 4.5 (2.4)
Statistical Analysis 1: Comparison: Methadone HCl 0.3 mg/kg vs Methadone HCl 0.4 mg/kg vs Control Group; Test type: Other — ANOVA; p = .962, ANOVA; F statistic = .962

3. Secondary Outcome: Cmax of R and S Methadone
Description: Cmax is the maximum (or peak) serum concentration that a drug achieves in a specified compartment or test area of the body after the drug has been administrated and before the administration of a second dose.
Time Frame: 96 hours
Population: Methadone clearance was only measured in the two groups that received methadone
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Methadone HCl 0.3 mg/kg | Methadone HCl 0.4 mg/kg
Number analyzed (Participants) | 20 | 14
ng/ml
  R- Methadone | 97 (37) | 175 (93)
  S- Methadone | 127 (43) | 226 (113)

ADVERSE EVENTS:
Time Frame: Up to 6 days post-preoperative.
Description: Patients were assessed each day, in the morning, for events.
Arm/Group | Methadone HCl 0.3 mg/kg | Methadone HCl 0.4 mg/kg | Control Group
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/14 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/14 | 0/16
Other Adverse Events (participants affected / at risk) | 6/20 | 6/14 | 8/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Methadone HCl 0.3 mg/kg (N=20) | Methadone HCl 0.4 mg/kg (N=14) | Control Group (N=16)
Excessive sedation (Surgical and medical procedures) | 1 | 0 | 1
Respiratory Depression (Respiratory, thoracic and mediastinal disorders) | 4 | 6 | 7 — Respiratory Rate <8/min or Saturations <90% for more than 30 sec
Ileus (Gastrointestinal disorders) | 1 | 0 | 0 — Delayed return of bowel sounds

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2017-01-31): https://cdn.clinicaltrials.gov/large-docs/73/NCT01990573/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2014-09-10): https://cdn.clinicaltrials.gov/large-docs/73/NCT01990573/Prot_SAP_001.pdf